CLINICAL TRIAL: NCT01354197
Title: Multicenter Study of Outcome and Adverse Events in Surgical Intensive Care Unit of Thai University Hospital
Brief Title: The Thai Surgical Intensive Care Study (Thai-SICU Study)
Acronym: THAI-SICU
Status: Completed | Type: Observational
Sponsor: Royal College of Anesthesiologists of Thailand (Other)
Collaborators: Siriraj Hospital (Other); Chulalongkorn University (Other); Chiang Mai University (Other); Prince of Songkla University (Other); Khon Kaen University (Other); Srinakharinwirot University (Other); Royal Thai Army Medical Department (Other Government); Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government); Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 40-53-11
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Complications of Surgical and Medical Care: General Terms; Adverse Reaction to Drug; Sequelae of External Causes of Morbidity and Mortality; Critical Illness
Keywords: Adverse events; Mortality; Readmission; Surgical intensive care unit
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All ICU admission patients: All ICU admission to surgical intensive care unit at cohort time

SUMMARY:
The study observed the 28 days mortality of 9 participated University base surgical intensive care unit (SICU) as well as the occurrence of adverse events in SICU.

DETAILED DESCRIPTION:
The adverse events included pulmonary aspiration, pulmonary emboli, drug error, new stroke, symptomatic deep vein thrombosis, pneumothorax, unplanned extubation, upper GI hemorrhage, myocardial infarction, abdominal hypertension, acute lung injury(ALI)/acute respiratory distress syndrome (ARDS), re-intubation within 72 hours, delirium, cardiac arrest, new arrhythmia, acute kidney injury, sepsis

ELIGIBILITY:
Inclusion Criteria:

* All SICU admission patients

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All SICU admission patients
Sampling Method: Non-Probability Sample
Enrollment: 4652 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suneerat Kongsayreepong, MD.FRCAT, Study Chair — Mahidol University
Locations (9):
- Thailand (9):
  - Department of Surgery and Department of Anesthesiology, Bangkok metropolitan medical college and Vajira hospital, Bangkok, Bangkok
  - Department of Anesthesiology, Faculty of Medicine, Chulalongkorn hospital, Bangkok, Bangkok
  - Department of Anesthesiology, Faculty of Medicine, Ramathibodi hospital, Bangkok, Bangkok
  - Department of Surgery, Pramongkudklao hospital, Bangkok, Bangkok
  - Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Bangkok, Bangkok
  - Department of Surgery, Faculty of Medicine, Maharaj Nakorn Chiang Mai hospital, Chiang Mai, Chiang Mai
  - Department of Anesthesiology, Faculty of Medicine, Srinakarin hospital, Khon Kaen, Khon Khon
  - Department of Anesthesiology, Nakhon Nayok, Nakorn Nayok
  - Department of Surgery and Department of Anesthesiology, Songkhla, Songkha

IPD SHARING:
Plan to Share IPD: Yes
All the data was managed by the the Medical Research Network of the Consortium of Thai Medical Schools (MedResNet)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All ICU Admission Patients
Started | 4652
Completed | 4652
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Survive at Day 28: The patients who survived at 28 days after surgical ICU admission.
- Non-survive at Day 28: The patients who non-survived at 28 days after surgical ICU admission.
- Total: Total of all reporting groups
Arm/Group | Survive at Day 28 | Non-survive at Day 28 | Total
Number analyzed (Participants) | 4010 | 642 | 4652
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (17.3) | 63.7 (17.4) | 61.7 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1692 | 231 | 1923
  Male | 2318 | 411 | 2729
Race/Ethnicity, Customized [Number; unit: participants]
  Thai | 4010 | 642 | 4652
Region of Enrollment [Number; unit: participants]
  Thailand | 4010 | 642 | 4652

OUTCOME MEASURES:

1. Primary Outcome: Overall Mortality
Description: Number of Participants who Did Not Survive up to 28 days after surgical ICU admission
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | All ICU Admission Patients
Number analyzed (Participants) | 4652
participants | 642

2. Secondary Outcome: Readmission to ICU
Description: Number of Participants with Readmission to ICU up to 3 days (72 hours) after discharge from ICU
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | All ICU Admission Patients
Number analyzed (Participants) | 4652
participants | 144

ADVERSE EVENTS:
Time Frame: Up to 28 days after surgical ICU admission
Description: The adverse events were collected up to 28 days in all participants who survive at day 28 and did not survive at day 28 after surgical ICU admission
Groups:
- Survive at Day 28: Number of participants who survive at day 28
- Non-survive at Day 28: Number of participants who Did Not survive at day 28
Arm/Group | Survive at Day 28 | Non-survive at Day 28
Serious Adverse Events (participants affected / at risk) | 1070/4010 | 519/642
Other Adverse Events (participants affected / at risk) | 253/4010 | 90/642
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Survive at Day 28 (N=4010) | Non-survive at Day 28 (N=642)
Sepsis (Infections and infestations) | 607 (607) | 300 (300)
Cardiac arrest (Cardiac disorders) | 17 (17) | 209 (209)
Acute lung injury/ Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 119 (119) | 119 (119)
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
New arrhythmia (Cardiac disorders) | 184 (184) | 103 (103)
New stroke (Nervous system disorders) | 9 (9) | 2 (2)
Seizure (Nervous system disorders) | 26 (26) | 19 (19)
Myocardial infarction (Cardiac disorders) | 47 (47) | 19 (19)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 33 (33) | 22 (22)
Acute kidney injury (Renal and urinary disorders) | 491 (491) | 295 (295)
Intra-abdominal hypertension (Gastrointestinal disorders) | 54 (54) | 17 (17)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Survive at Day 28 (N=4010) | Non-survive at Day 28 (N=642)
Delirium (Nervous system disorders) | 117 (117) | 46 (46)
Reintubation within 72 hours (Respiratory, thoracic and mediastinal disorders) | 112 (112) | 29 (29)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 11 (11)
Unplanned extubation (Respiratory, thoracic and mediastinal disorders) | 41 (41) | 16 (16)
Self reported medication error (Surgical and medical procedures) | 7 (7) | 3 (3)
Pulmonary aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Symptomatic deep venous thrombosis (Vascular disorders) | 10 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No